CLINICAL TRIAL: NCT07026578
Title: Unravelling the Role of Apoptosis in Platelets Biogenesis Through the Study of the CYCS Mut-associated Thrombocytopenia THC4
Brief Title: Unravelling the Role of Apoptosis in Platelets Biogenesis Through the Study of the Thrombocytopenia THC4
Acronym: THC4
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Serena Barozzi, Biologist, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: THC4
Record Dates: First submitted 2025-03-13; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-04

CONDITIONS: Thrombocytopenia, Isolated; Thrombocytopenia 4; CYCS MUTATION- ASSOCIATED THROMBOCYTOPENIA THC4
Keywords: Apoptosis; Platelet biogenesis; Thrombocytopenia 4
MeSH Terms: conditions — Thrombocytopenia; Thrombocytopenia 4 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 25 mL of peripheral whole blood anticoagulated with ACD for platelet isolation and for separation of hematopoietic progenitors to differentiate megakaryocytes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CYCS mutated
  Interventions: Procedure: Blood draw for the laboratory assessment
- healthy controls
  Interventions: Procedure: Blood draw for the laboratory assessment

INTERVENTIONS:
Procedure: Blood draw for the laboratory assessment — This is an observational study . The procedures will be carried out in according to clinical practice

SUMMARY:
Inherited thrombocytopenias (ITs) are disorders characterized by a reduced platelet count, caused by variants in at least 40 genes. Mutations in CYCS cause a rare autosomal-dominant IT, named Thrombocytopenia 4 (THC4). The CYCS gene encodes cytochrome C (CytC), a small heme protein localized in mitochondria. It functions as an electron carrier in the respiratory chain as well as one of the main actors of the intrinsic pathway of apoptosis.

Although THC4 is the only disease associated with CYCS mutations, its clinical and molecular features are still poorly characterized. Moreover, pathogenesis of THC4 is still unclear. In vitro studies demonstrated that CYCS mutations exert a proapoptotic activity and enhanced peroxidase activity, as well as affect the mitochondrial respiratory function in yeast.

The role of apoptosis in platelet biogenesis is a highly controversial issue. Some studies suggested that megakaryocytes must undergo apoptosis to promote platelet release. In fact, mice carrying mutations impairing apoptosis exhibited thrombocytopenia and pharmacological inhibition of caspases blocked platelet production, supporting this hypothesis. Conversely, investigations on mice genetically modified for the BCL-2 family proteins, initiators of apoptosis, concluded that megakaryocytes must restrain apoptosis in order to generate platelets.

Since thrombocytopenia is the only phenotypic manifestation of CYCS mutations, the investigators believe that THC4 represents a unique model for deciphering the role of Cytc and apoptosis in megakaryopoiesis and platelet biogenesis.

Preliminary data:

The applicant unit is a reference center for ITs. The database includes 375 families; among these, 7 presented with mutations in CYCS gene, accounting for 26 THC4 patients.

Patients presented mild thrombocytopenia, normal mean platelet volume and morphology, without hematological or extra-hematological defects.

The investigators isolated platelets and hematopoietic progenitors from peripheral blood of 9 patients. Platelets were analyzed under baseline conditions; a part was treated with an inducer of apoptosis (ABT-737).

Surprisingly, the expression of cytC was found reduced in platelets of all analyzed patients. Platelets showed no signs of early death. Instead, when stimulated with ABT-737, they showed inability to undergo apoptosis, suggesting that CYCS mutations confer resistance to apoptosis.

Hematopoietic progenitors from 3 patients were differentiated in megakaryocytes. Maturation and differentiation were comparable between THC4 and healthy controls. Instead, their capability to form proplatelets was profoundly defective.

These preliminary data suggest that CytC deficit could be associated with inability to form proplatelets in THC4 megakaryocytes, and that this defect underlies thrombocytopenia, supporting the crucial role of cytC in platelet production.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of THC4, through the identification of a pathogenic variant of the CYCS gene
* Acquisition of written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with suspected Inherited Thrombocytopenia (IT) observed at the SC Medicina generale 1, Fondazione IRCCS Policlinico San Matteo
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathogenetic CYCS variants result in defective Cytc expression | The primary endpoint measurement will be performed immediately after the enrollment (baseline).
  The primary outcome of the study is to demonstrate that mutations in CYCS results in reduction of the expression of Cytochrome C in THC4 platelets. The primary endpoint will compare Cytochrome C expression in platelets between THC4 patients and healthy controls. This will be assessed by measuring Cytochrome C protein levels in platelet lysates collected from both groups. Western blotting will be used to quantify the amount of Cytochrome C protein.

SECONDARY OUTCOMES:
The impact of Cytochrome C (CytC) deficiency on apoptotic mechanisms evaluated as the comparison of the apoptotic markers between CYCS-silenced cells and cells transduced with the vector alone | The production of in vitro models and execution of tests to evaluate the apoptotic profile will take 2 weeks
  Once CytC deficiency has been confirmed, in vitro models will be created to study the effects on the apoptotic machinery. Parameters will be analyzed in CYCS-silenced cells and baseline cells in the presence or absence of apoptosis inducers: phosphatidylserine exposure, cell viability, depolarization of mitochondrial membranes. Extrinsic and intrinsic apoptotic pathways will be analyzed as the activation of initiator and executioner caspases with different techniques such as flow cytometry, immunofluorescence staining, and immunoblotting. All these results will be expressed as the percentage of positive cells after treatment with an apoptotic inducer relative to treated baseline cells. The data will be aggregated to determine if CytC deficiency results in an increased or decreased apoptotic rate in THC4, expressed as a higher or lower percentage of apoptotic cells in the absence of CytC.

OTHER OUTCOMES:
The effects of alterations of apoptotic mechanisms on megakaryopoiesis and platelet production evaluated as a decrease in CD61+ and CD42b+ cells and reduced ability to form proplatelets in vitro | Along with the measurement of Cytochrome C in platelets, circulating progenitors will be collected from patients, from which megakaryocytes will be differentiated in vitro, either immediately upon enrollment (baseline)
  The investigators will assess the following:
  1. Megakaryocyte differentiation (% CD61 expression).
  2. Megakaryocyte maturation (co-expression % of CD61 or CD41/CD42b and ploidy).
  3. Formation of proplatelet extensions, either in suspension or upon adhesion to proteins of the bone marrow extracellular matrix (% of proplatelet-bearing cells).
  All these results will be expressed as the percentage of positive megakaryocytes from THC4 patients compared to those from healthy controls. These data will be aggregated to conclude if CytC deficiency causes defects in megakaryopoiesis in THC4.

CONTACTS AND LOCATIONS:
Locations (1):
- SC Medicina Generale 1, Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy